CLINICAL TRIAL: NCT01916213
Title: The Valve of Hyaluronic Binding Selection (PICSI) in Improving IVF Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 12-065
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2014-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PICSI (Active Comparator): PICSI dish ( MidAtlantic Diagnostics Inc) has been developed to select the specific sperm to be used for the ICSI procedure using the same principles as the Sperm Hyaluronan Binding Assay. HA-mediated ICSI sperm selection( PICSI) uses Falcon Petri dishes that feature three microdots of hyaluronan hydrogel attached to the interior bottom: mature, biochemically competent spermatozoa bind to hyaluronan, where they can be isolated and used for ICSI
  Interventions: Procedure: PICSI
- ICSI (Active Comparator)
  Interventions: Procedure: PICSI

INTERVENTIONS:
Procedure: PICSI — If the oocytes are randomized to ICSI during the retrieval they will be ordered by the 1,4,5 8th best oocyte and PICSI to the 2,3, 6 7th best oocytes or the reverse if PICSI is selected. If one cohort is superior that cohort should be chosen by the blinded physician and the alternate cohort frozen or discarded based on their quality. This will ensure that the couple will always have the opportunity to have good quality embryo transferred regardless of how they are randomized. If there are no good quality embryos in the selected cycle we will consider it a failed transfer for that cycle and we will transfer the good quality embryos from the non- selected group as a fresh embryo transfer. For example if a couple is randomized to ICSI and all the ICSI embryos are poor quality but the PICSI embryos are good quality we will consider it a failed ICSI transfer and transfer the PICSI embryos as a fresh embryo transfer.
  Other Names: The PICSI® dish is based on the research documenting that mature and structurally sound sperm will bind to hyaluronan.; CE marked (CE 0120)

SUMMARY:
The investigators would like to assess whether selecting mature sperm using PICSI (selecting for sperm that bind hyaluronan) can optimize the IVF outcome of ICSI .

Aim

1. Primary outcome: To compare routine sperm selection using ICSI with sperm selection using PICSI plates in terms of implantation and fertilization rates for couples with male factor fertility
2. Secondary outcome : To compare live birth rates ,ongoing pregnancies and miscarriage rates for couples with male factor infertility using routine sperm selection with ICSI compared to using PICSI plates for sperm selection

Hypothesis:

Sperm selected for ICSI using (PICSI) will reveal increased implantation rates in comparison to sperm selected for conventional ICSI

ELIGIBILITY:
Inclusion Criteria:

* In order to participate in the study women must be 42 years old or younger and suffer from male factor infertility however they may have other causes for their infertility
* male factor infertility as defined by one or more of the following sperm parameters: <20 Million /ml sperm concentration < 30% normal morphology < 3% Kruger morphology < 50% motility sion Criteria:

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
implantation rate | 12 months

SECONDARY OUTCOMES:
fertilization rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Continuum Reproductive Center, New York, New York, United States